CLINICAL TRIAL: NCT05491577
Title: Factors Associated With Quality of Life Outcomes in Diabetic Patients With Chronic Wound-free Charcot Foot
Brief Title: Factors Associated With an Evolution in the Quality of Life of Diabetic Patients With Chronic, Wound-free Charcot Foot
Acronym: CHARQUAM
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: SI RIPH 2G : 22.01571.000083
Record Dates: First submitted 2022-07-29; First posted 2022-08-08 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Charcot Joint of Foot; Osteoarthropathy
Keywords: Diabetes complications; Diabetic foot; Osteoarthropathy
MeSH Terms: conditions — Diabetes Complications; Diabetic Foot | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Filling in the SF-36, FAAM-F, PHQ-9, PHQ-2 and the simplified version of the EPICES score questionnaire — The SF-36, FAAM-F, PHQ-9, PHQ-2 and the simplified version of the EPICES score questionnaire will all be filled in by the patients.

SUMMARY:
Charcot foot, characterized by progressive destructive damage to bone, soft tissue and tendons, involving joint dislocation in the ankle and foot, is a complication of diabetes that is still poorly understood by patients and caregivers. The clinical signs are non-specific and it is therefore largely underestimated due to a delay in diagnosis/lack of diagnosis.This study will be on a prospective multicenter cohort of patients with chronic Charcot's foot in France to evaluate the evolution of quality of life at 2 years, as well as predictive factors in order to better identify subjects with the worst outcome among this population.

Our hypothesis is that, in patients with chronic Charcot foot, the deterioration in quality of life over time is primarily related to loss of foot and ankle functionality, foot and ankle deformity and the presence of foot wounds/comorbidities/severe diabetic complications.

DETAILED DESCRIPTION:
Diabetes mellitus is a chronic disease, representing a major public health problem. An estimated 537 million people have diabetes. Charcot foot, also known as neurogenic osteoarthropathy (NAO), is one of the complications of diabetes secondary to diabetic neuropathy. It is characterized by progressive destructive damage to bone, soft tissue and tendons, involving joint dislocation in the ankle and foot. Charcot foot is a complication of diabetes that is still poorly understood by patients and caregivers, with non-specific clinical signs. It is therefore largely underestimated, since it is estimated that there is a delay in diagnosis or a lack of diagnosis in approximately 25% of cases.

The objective of our study is to conduct a prospective multicenter cohort of patients with chronic Charcot's foot in France in order to evaluate the evolution of the quality of life at 2 years, as well as its predictive factors. In this way, we will be better able to identify the subjects with the worst outcome among the chronic Charcot foot population.

Our hypothesis is that the deterioration in quality of life over time in patients with chronic Charcot foot is primarily related to loss of foot and ankle functionality, foot and ankle deformity, the presence of foot wounds and/or comorbidities or severe diabetic complications.

ELIGIBILITY:
Inclusion Criteria:

* patients with Type 1 or 2 diabetes or secondary diabetes
* patient hospitalized or consulting for osteoarthropathy in its chronic stage, without wounds
* patients affiliated to or beneficiaries of a health insurance scheme.
* adult patients (≥18 years old).

Exclusion Criteria:

* patients with non-diabetic osteoarthropathy of the nerves.
* patients with acute diabetic osteoarthropathy of the nerves.
* patients with a foot ulcer
* patients who have expressed opposition to participating in the study.
* patients in an exclusion period determined by another study.
* patients under court protection, guardianship or trusteeship.
* patients for whom it is impossible to give informed information.
* pregnant, parturient, or breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population corresponds to all diabetic patients (Type 1, 2 or secondary diabetes) hospitalized or consulting for chronic diabetic osteoarthropathy of the nerves, without wound managed in the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2028-01-22 (Estimated)

PRIMARY OUTCOMES:
Results of the SF36 questionnaire at inclusion | Day 0
  The SF-36 questionnaire is a quality of life questionnaire that includes 36 questions divided into 8 different categories (physical functioning, limitations due to physical condition, physical pain, perceived health, vitality, social functioning or well-being, limitations due to mental condition, mental health). These 8 dimensions are used to calculate two scores on the quality of life of individuals: the physical composite score and the mental composite score. The higher the score, the greater the capacity. It is self-administered and takes less than 10 minutes. Higher scores indicate better quality of life. The French version has been validated and has satisfactory psychometric properties. Score from 0 to 100.
Results of the FAAM-F questionnaire at inclusion | Day 0
  The FAAM is a self-administered questionnaire that measures physical function of the foot and ankle. It is adapted and validated in the evaluation of diabetic foot disease. It consists of an assessment of activity of daily living and a sports assessment. The FAAM has been translated and validated in French. Score from 0 to 100.
Results of the SF36 questionnaire at Month 12 | Month 12
  The SF-36 questionnaire is a quality of life questionnaire that includes 36 questions divided into 8 different categories (physical functioning, limitations due to physical condition, physical pain, perceived health, vitality, social functioning or well-being, limitations due to mental condition, mental health). These 8 dimensions are used to calculate two scores on the quality of life of individuals: the physical composite score and the mental composite score. The higher the score, the greater the capacity. It is self-administered and takes less than 10 minutes. Higher scores indicate better quality of life. The French version has been validated and has satisfactory psychometric properties. Score from 0 to 100.
Results of the FAAM-F questionnaire at Month 12 | Month 12
  The FAAM is a self-administered questionnaire that measures physical function of the foot and ankle. It is adapted and validated in the evaluation of diabetic foot disease. It consists of an assessment of activity of daily living and a sports assessment. The FAAM has been translated and validated in French. Score from 0 to 100.
Results of the SF36 questionnaire at Month 24 | Month 24
  The SF-36 questionnaire is a quality of life questionnaire that includes 36 questions divided into 8 different categories (physical functioning, limitations due to physical condition, physical pain, perceived health, vitality, social functioning or well-being, limitations due to mental condition, mental health). These 8 dimensions are used to calculate two scores on the quality of life of individuals: the physical composite score and the mental composite score. The higher the score, the greater the capacity. It is self-administered and takes less than 10 minutes. Higher scores indicate better quality of life. The French version has been validated and has satisfactory psychometric properties. Score from 0 to 100.
Results of the FAAM-F questionnaire at Month 24 | Month 24
  The FAAM is a self-administered questionnaire that measures physical function of the foot and ankle. It is adapted and validated in the evaluation of diabetic foot disease. It consists of an assessment of activity of daily living and a sports assessment. The FAAM has been translated and validated in French. Score from 0 to 100.

SECONDARY OUTCOMES:
A. Evolution of X-ray measurements of bone and joint deformity of the foot. Lisfranc metatarsal misalignment (Méary's Line) | Day 0
  In normal metatarsal alignment, the lateral border of the 1st metatarsal is aligned with lateral border of 1st (medial) cuneiform. The medial border of 2nd metatarsal is aligned with the medial border of 2nd (intermediate) cuneiform.The medial border of the 3rd (lateral) cuneiform should align with the medial border of the 3rd metatarsal. The lateral border of the 3rd (lateral) cuneiform should align with the lateral border of the 3rd metatarsal. The medial border of the 4th metatarsal is aligned with the medial border of the cuboid. The lateral margin of the 5th metatarsal can project lateral to cuboid by up to 3 mm on oblique. This alignment is known as the Méary Line and is assessed in front view.
A. Evolution of X-ray measurements of bone and joint deformity of the foot. Lisfranc metatarsal misalignment (Méary's Line) | Month 12
  In normal metatarsal alignment, the lateral border of the 1st metatarsal is aligned with lateral border of 1st (medial) cuneiform. The medial border of 2nd metatarsal is aligned with the medial border of 2nd (intermediate) cuneiform.The medial border of the 3rd (lateral) cuneiform should align with the medial border of the 3rd metatarsal. The lateral border of the 3rd (lateral) cuneiform should align with the lateral border of the 3rd metatarsal. The medial border of the 4th metatarsal is aligned with the medial border of the cuboid. The lateral margin of the 5th metatarsal can project lateral to cuboid by up to 3 mm on oblique. This alignment is known as the Méary Line and is assessed in front view.
A. Evolution of X-ray measurements of bone and joint deformity of the foot. Lisfranc metatarsal misalignment (Méary's Line) | Month 24
  In normal metatarsal alignment, the lateral border of the 1st metatarsal is aligned with lateral border of 1st (medial) cuneiform. The medial border of 2nd metatarsal is aligned with the medial border of 2nd (intermediate) cuneiform.The medial border of the 3rd (lateral) cuneiform should align with the medial border of the 3rd metatarsal. The lateral border of the 3rd (lateral) cuneiform should align with the lateral border of the 3rd metatarsal. The medial border of the 4th metatarsal is aligned with the medial border of the cuboid. The lateral margin of the 5th metatarsal can project lateral to cuboid by up to 3 mm on oblique. This alignment is known as the Méary Line and is assessed in front view.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot: Méary's angle. | Day 0
  Meary's angle (the angle between the line from the center of the talus body, intersecting the neck and head of the talus, and the line through the longitudinal axis of the 1st metatarsal) will be measured in profile view, in degrees. The normal value is about 0°.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot: Méary's angle. | Month 12
  Meary's angle (the angle between the line from the center of the talus body, intersecting the neck and head of the talus, and the line through the longitudinal axis of the 1st metatarsal) will be measured in profile view, in degrees. The normal value is about 0°.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot: Méary's angle. | Month 24
  Meary's angle (the angle between the line from the center of the talus body, intersecting the neck and head of the talus, and the line through the longitudinal axis of the 1st metatarsal) will be measured in profile view, in degrees. The normal value is about 0°.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Calcaneal slope | Day 0
  The calcaneal slope angle (line tangent to the inferior cortex of the calcaneus (angle between this line and a horizontal line) will be measured in degrees. Normal values are10-30° on the profile X-ray.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Calcaneal slope | Month 12
  The calcaneal slope angle (line tangent to the inferior cortex of the calcaneus (angle between this line and a horizontal line) will be measured in degrees. Normal values are10-30° on the profile X-ray.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Calcaneal slope | Month 24
  The calcaneal slope angle (line tangent to the inferior cortex of the calcaneus (angle between this line and a horizontal line) will be measured in degrees. Normal values are10-30° on the profile X-ray.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Djian Annonier angle | Day 0
  The Djian-Annonier angle will be measured (line between lower point of the talo-navicular joint and lower point of the medial sesamoid bone at the hallux). Line tangent to the inferior surface of the calcaneus. Normal value: 120-130° on profile X-ray.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Djian Annonier angle | Month 12
  The Djian-Annonier angle will be measured (line between lower point of the talo-navicular joint and lower point of the medial sesamoid bone at the hallux). Line tangent to the inferior surface of the calcaneus. Normal value: 120-130° on profile X-ray.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Djian Annonier angle | Month 24
  The Djian-Annonier angle will be measured (line between lower point of the talo-navicular joint and lower point of the medial sesamoid bone at the hallux). Line tangent to the inferior surface of the calcaneus. Normal value: 120-130° on profile X-ray.
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Rearfoot alignment | Day 0
  The rearfoot alignment angle i.e. angle between the axis of the tibia and the line between the middle of the plantar support plane and the middle of talus will be measured in degrees..
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Rearfoot alignment | Month 12
  The rearfoot alignment angle i.e. angle between the axis of the tibia and the line between the middle of the plantar support plane and the middle of talus will be measured in degrees..
A. Evolution of the radiologic measurements of bone and joint deformity of the foot. Rearfoot alignment | Month 24
  The rearfoot alignment angle i.e. angle between the axis of the tibia and the line between the middle of the plantar support plane and the middle of talus will be measured in degrees..
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Retinopathy | Month 24
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Retinopathy | Month 12
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Peripheral vegetative neuropathy. | Day 0
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Peripheral vegetative neuropathy. | Month 12
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Peripheral vegetative neuropathy. | Month 24
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Nephropathy. | Day 0
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Nephropathy. | Month 12
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Nephropathy. | Month 24
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Lower extremity arteriopathy | Day 0
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Lower extremity arteriopathy | Month 12
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Lower extremity arteriopathy | Month 24
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Supra-aortic trunk involvement | Day 0
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Supra-aortic trunk involvement | Month 12
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Supra-aortic trunk involvement | Month 24
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Coronary artery disease | Day 0
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Coronary artery disease | Month 12
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Coronary artery disease | Month 24
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Heart failure | Day 0
  YES/NO (measured according to a Left Ventricle Ejection Fraction of less than 50%)
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Heart failure | Month 12
  YES/NO (measured according to a Left Ventricle Ejection Fraction of less than 50%)
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Heart failure | Month 24
  YES/NO (measured according to a Left Ventricle Ejection Fraction of less than 50%)
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. History of strokes | Day 0
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. History of strokes | Month 12
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. History of strokes | Month 24
  YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Arterial hypertension | Day 0
  Pressure over 140/90mmHg : YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Arterial hypertension | Month 12
  Pressure over 140/90mmHg : YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Arterial hypertension | Month 24
  Pressure over 140/90mmHg : YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Smoking | Day 0
  Does the patient smoke : YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Smoking | Month 12
  Does the patient smoke : YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Smoking | Month 24
  Does the patient smoke : YES/NO
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Alcohol status | Day 0
  Does the patient drink more than 3 glasses of alcohol per day : YES/NO alcohol status Charlson score
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Alcohol status | Month 12
  Does the patient drink more than 3 glasses of alcohol per day : YES/NO alcohol status Charlson score
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Alcohol status | Month 24
  Does the patient drink more than 3 glasses of alcohol per day : YES/NO alcohol status Charlson score
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Charlson Comorbidity Index | Day 0
  The Charlson comorbidity index predicts the 1-year mortality for patient with a range of comorbid conditions, e.g. heart disease, AIDS, or cancer (a total of 22 conditions). Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. Scores are summed to provide a total score to predict mortality. Clinical conditions and associated scores are as follows:
  1. each: Myocardial infarct, congestive heart failure, peripheral vascular disease, dementia, cerebrovascular disease, chronic lung disease, connective tissue disease, ulcer, chronic liver disease, diabetes.
  2. each: Hemiplegia, moderate or severe kidney disease, diabetes with end organ damage, tumor, leukemia, lymphoma.
  3. each: Moderate or severe liver disease.
  6 each: Malignant tumor, metastasis, AIDS.
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Charlson Comorbidity Index | Month 12
  The Charlson comorbidity index predicts the 1-year mortality for patient with a range of comorbid conditions, e.g. heart disease, AIDS, or cancer (a total of 22 conditions). Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. Scores are summed to provide a total score to predict mortality. Clinical conditions and associated scores are as follows:
  1. each: Myocardial infarct, congestive heart failure, peripheral vascular disease, dementia, cerebrovascular disease, chronic lung disease, connective tissue disease, ulcer, chronic liver disease, diabetes.
  2. each: Hemiplegia, moderate or severe kidney disease, diabetes with end organ damage, tumor, leukemia, lymphoma.
  3. each: Moderate or severe liver disease.
  6 each: Malignant tumor, metastasis, AIDS.
B. Estimated prevalence of complications of diabetes and comorbidities at inclusion. Charlson Comorbidity Index | Month 24
  The Charlson comorbidity index predicts the 1-year mortality for patient with a range of comorbid conditions, e.g. heart disease, AIDS, or cancer (a total of 22 conditions). Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. Scores are summed to provide a total score to predict mortality. Clinical conditions and associated scores are as follows:
  1. each: Myocardial infarct, congestive heart failure, peripheral vascular disease, dementia, cerebrovascular disease, chronic lung disease, connective tissue disease, ulcer, chronic liver disease, diabetes.
  2. each: Hemiplegia, moderate or severe kidney disease, diabetes with end organ damage, tumor, leukemia, lymphoma.
  3. each: Moderate or severe liver disease.
  6 each: Malignant tumor, metastasis, AIDS.
C. Medical and/or surgical treatment for Charcot foot. | Day 0
  All medical and/or surgical treatment for Charcot foot will be recorded.
C. Medical and/or surgical treatment for Charcot foot. | Month 12
  All medical and/or surgical treatment for Charcot foot will be recorded.
C. Medical and/or surgical treatment for Charcot foot. | Month 24
  All medical and/or surgical treatment for Charcot foot will be recorded.
D. Incidence of hospitalization | Month 12
  The number of hospitalizations (if any) will be noted.
D. Incidence of hospitalization | Month 24
  The number of hospitalizations (if any) will be noted.
E. Presence of a wound/wounds | Month 12
  YES/NO and number thereof.
E. Presence of a wound/wounds | Month 24
  YES/NO and number thereof.
E. Presence of an infection | Month 12
  YES/NO
E. Presence of an infection | Month 24
  YES/NO
F. Presence of an amputation at inclusion | Day 0
  YES/NO (or, if planned, time to amputation in days).
G. Estimated incidence of amputations | Month 12
  YES/NO (or, if planned, time to amputation in days).
G. Presence of an amputation | Month 24
  YES/NO (or, if planned, time to amputation in days).
H. Precarity of patients with chronic Charcot foot. | Day 0
  The EPICES (Evaluation de la précarité et des inégalités de santé dans les Centres d'examens) score is an individual indicator of precariousness that takes into account the multidimensional nature of precariousness. The main interest of the EPICES score is to capture populations which, while not covered by traditional administrative indicators of precariousness present the same health risks. A threshold of 30 is considered as precariousness according to EPICES.
H. Precarity of patients with chronic Charcot foot. | Month 12
  The EPICES (Evaluation de la précarité et des inégalités de santé dans les Centres d'examens) score is an individual indicator of precariousness that takes into account the multidimensional nature of precariousness. The main interest of the EPICES score is to capture populations which, while not covered by traditional administrative indicators of precariousness present the same health risks. A threshold of 30 is considered as precariousness according to EPICES.
H. Precarity of patients with chronic Charcot foot. | Month 24
  The EPICES (Evaluation de la précarité et des inégalités de santé dans les Centres d'examens) score is an individual indicator of precariousness that takes into account the multidimensional nature of precariousness. The main interest of the EPICES score is to capture populations which, while not covered by traditional administrative indicators of precariousness present the same health risks. A threshold of 30 is considered as precariousness according to EPICES.
I. Depression according to the PHQ-2 self-questionnaire | Day 0
  The purpose of the PHQ-2 is to screen for depression in a "first-step" approach. there are 2 questions referring to the patient's feelings over the previous 2 weeks ( 0 = Not at all and 3 = Nearly every day). A PHQ-2 score ranges from 0-6 and a score of 3 is the optimal cutoff point when using the PHQ-2 to screen for depression. If the score is 3 or greater, major depressive disorder is likely and the PHQ-9 questionnaire should then be used.
I. Depression according to the PHQ-2 self-questionnaire | Month 24
  The purpose of the PHQ-2 is to screen for depression in a "first-step" approach. there are 2 questions referring to the patient's feelings over the previous 2 weeks ( 0 = Not at all and 3 = Nearly every day). A PHQ-2 score ranges from 0-6 and a score of 3 is the optimal cutoff point when using the PHQ-2 to screen for depression. If the score is 3 or greater, major depressive disorder is likely and the PHQ-9 questionnaire should then be used.
I. Depression according to the PHQ-2 self-questionnaire | Month 12
  The purpose of the PHQ-2 is to screen for depression in a "first-step" approach. there are 2 questions referring to the patient's feelings over the previous 2 weeks ( 0 = Not at all and 3 = Nearly every day). A PHQ-2 score ranges from 0-6 and a score of 3 is the optimal cutoff point when using the PHQ-2 to screen for depression. If the score is 3 or greater, major depressive disorder is likely and the PHQ-9 questionnaire should then be used.
I. Depression according to the PHQ-9 self-questionnaire | Day 0
  The PHQ-9 questionnaire is a set of 9 questions referring to the patients feelings over the previous 2 weeks with answers ranging from 0 = Not at all to 3 = Nearly every day. Interpreted as follows : 1-4 = minimum depression ; 5-9 = slight depression;10-14 = moderate depression;15-19 = moderately severe depression and 20-27 = severe depression.
I. Depression according to the PHQ-9 self-questionnaire | Month 12
  The PHQ-9 questionnaire is a set of 9 questions referring to the patients feelings over the previous 2 weeks with answers ranging from 0 = Not at all to 3 = Nearly every day. Interpreted as follows : 1-4 = minimum depression ; 5-9 = slight depression;10-14 = moderate depression;15-19 = moderately severe depression and 20-27 = severe depression.
I. Depression according to the PHQ-9 self-questionnaire | Month 24
  The PHQ-9 questionnaire is a set of 9 questions referring to the patients feelings over the previous 2 weeks with answers ranging from 0 = Not at all to 3 = Nearly every day. Interpreted as follows : 1-4 = minimum depression ; 5-9 = slight depression;10-14 = moderate depression;15-19 = moderately severe depression and 20-27 = severe depression.
J. Mortality rate | Month 12
  Vital status (dead/alive)
J. Mortality rate | Month 24
  Vital status (dead/alive)
K. Sanders Classification of the Charcot Foot | Day 0
  The Sanders classification will be used to assess the degree of damage to the patient's foot as follows :
  Sanders I = Metatarsophalangeal involvement (forefoot) Sanders II= Tarsometatarsal joint involvement Sanders III= Tarsal joints involvement Sanders IV= Ankle involvement Sanders V= Posterior calcaneus involvement (tuberosity of the calcaneus, avulsion of the Achilles tendon)
  and all information will be recorded for the evaluation of the patient's quality of life.
K. Sanders Classification of the Charcot Foot | Month 12
  The Sanders classification will be used to assess the degree of damage to the patient's foot as follows :
  Sanders I = Metatarsophalangeal involvement (forefoot) Sanders II= Tarsometatarsal joint involvement Sanders III= Tarsal joints involvement Sanders IV= Ankle involvement Sanders V= Posterior calcaneus involvement (tuberosity of the calcaneus, avulsion of the Achilles tendon)
  and all information will be recorded for the evaluation of the patient's quality of life.

OTHER OUTCOMES:
Sex of patients | Day 0
  MALE/FEMALE
Age of patients | Day 0
  In years
Patient's personal situation | Day 0
  Lives alone/ Lives with family or has family nearby/Primary caregiver of another person/Lives in a bungalow/ Lives in a 2 or 3-storey house/ No fixed abode / Visits from a state-registered nurse/ Home help / Physiotherapy
Patient's personal situation | Month 12
  Lives alone/ Lives with family or has family nearby/Primary caregiver of another person/Lives in a bungalow/ Lives in a 2 or 3-storey house/ No fixed abode / Visits from a state-registered nurse/ Home help / Physiotherapy
Patient's personal situation | Month 24
  Lives alone/ Lives with family or has family nearby/Primary caregiver of another person/Lives in a bungalow/ Lives in a 2 or 3-storey house/ No fixed abode / Visits from a state-registered nurse/ Home help / Physiotherapy
Patient's level of education | Day 0
  The patient's level of education will be recorded:
  No diploma (including: no schooling or schooling completed before the end of elementary school; schooling completed until the end of elementary school or completed before the end of junior high school; schooling until the end of junior high school or beyond)
  * Primary school certificate;
  * BEPC, brevet élémentaire, brevet des collèges, DNB ;
  * CAP, BEP or equivalent diploma;
  * Baccalaureate, vocational diploma including: general or technological baccalaureate, higher diploma, capacity in law, DAEU, ESEU; vocational baccalaureate, vocational, technician or teaching diploma, equivalent diploma;
  * BTS, DUT, DEUG, DEUST, health or social diploma of Bac+2 level, equivalent diploma;
  * Bachelor's degree, professional license, master's degree, equivalent diploma of bac+3 or bac+4 level;
  * Master's degree, DEA, DESS, diploma from an engineering school at Bac+5 level, health doctorate;
  * Research doctorate (not in health).
Patient's level of education | Month 12
  The patient's level of education will be recorded:
  No diploma (including: no schooling or schooling completed before the end of elementary school; schooling completed until the end of elementary school or completed before the end of junior high school; schooling until the end of junior high school or beyond)
  * Primary school certificate;
  * BEPC, brevet élémentaire, brevet des collèges, DNB ;
  * CAP, BEP or equivalent diploma;
  * Baccalaureate, vocational diploma including: general or technological baccalaureate, higher diploma, capacity in law, DAEU, ESEU; vocational baccalaureate, vocational, technician or teaching diploma, equivalent diploma;
  * BTS, DUT, DEUG, DEUST, health or social diploma of Bac+2 level, equivalent diploma;
  * Bachelor's degree, professional license, master's degree, equivalent diploma of bac+3 or bac+4 level;
  * Master's degree, DEA, DESS, diploma from an engineering school at Bac+5 level, health doctorate;
  * Research doctorate (not in health).
Patient's level of education | Month 24
  The patient's level of education will be recorded:
  No diploma (including: no schooling or schooling completed before the end of elementary school; schooling completed until the end of elementary school or completed before the end of junior high school; schooling until the end of junior high school or beyond)
  * Primary school certificate;
  * BEPC, brevet élémentaire, brevet des collèges, DNB ;
  * CAP, BEP or equivalent diploma;
  * Baccalaureate, vocational diploma including: general or technological baccalaureate, higher diploma, capacity in law, DAEU, ESEU; vocational baccalaureate, vocational, technician or teaching diploma, equivalent diploma;
  * BTS, DUT, DEUG, DEUST, health or social diploma of Bac+2 level, equivalent diploma;
  * Bachelor's degree, professional license, master's degree, equivalent diploma of bac+3 or bac+4 level;
  * Master's degree, DEA, DESS, diploma from an engineering school at Bac+5 level, health doctorate;
  * Research doctorate (not in health).
Patient's professional activity | Day 0
  The patient's professional activity (if any) will be recorded
Patient's professional activity | Month 12
  The patient's professional activity (if any) will be recorded
Patient's professional activity | Month 24
  The patient's professional activity (if any) will be recorded
Nature of diabetes | Day 0
  The nature of the patient's diabetes will be recorded (Type 1, Type 2, unknown, other).
Nature of diabetes | Month 12
  The nature of the patient's diabetes will be recorded (Type 1, Type 2, unknown, other).
Nature of diabetes | Month 24
  The nature of the patient's diabetes will be recorded (Type 1, Type 2, unknown, other).
Age of diabetes | Day 0
  The age of the patient's diabetes will be recorded (More than 20 years/ 10 to 20 years/ 5 to 10 years/ less than 5 years/ unknown).
Age of diabetes | Month 12
  The age of the patient's diabetes will be recorded (More than 20 years/ 10 to 20 years/ 5 to 10 years/ less than 5 years/ unknown).
Age of diabetes | Month 24
  The age of the patient's diabetes will be recorded (More than 20 years/ 10 to 20 years/ 5 to 10 years/ less than 5 years/ unknown).
Presence of other complications: Retinopathy | Day 0
  YES/NO
Presence of other complications: Retinopathy | Month 12
  YES/NO
Presence of other complications: Retinopathy | Month 24
  YES/NO
Presence of other complications: decreased visual acuity | Day 0
  YES/NO
Presence of other complications: decreased visual acuity | Month 12
  YES/NO
Presence of other complications: decreased visual acuity | Month 24
  YES/NO
Presence of other complications: Nephropathy | Day 0
  YES/NO and the nature thereof (Insipid nephropathy / Proteinuric nephropathy / Chronic kidney failure)
Presence of other complications: Nephropathy | Month 12
  YES/NO and the nature thereof (Insipid nephropathy / Proteinuric nephropathy / Chronic kidney failure)
Presence of other complications: Nephropathy | Month 24
  YES/NO and the nature thereof (Insipid nephropathy / Proteinuric nephropathy / Chronic kidney failure)
Presence of other complications: Abnormal glomerular filtration rate (GFR) | Day 0
  GFR between 60 and 89ml/min/1.73 m² / GFR between 15 and 29ml/min/1.73 m² / GFR < 15 ml/min/1.73 m²
Presence of other complications: Abnormal glomerular filtration rate (GFR) | Month 12
  GFR between 60 and 89ml/min/1.73 m² / GFR between 15 and 29ml/min/1.73 m² / GFR < 15 ml/min/1.73 m²
Presence of other complications: Abnormal glomerular filtration rate (GFR) | Month 24
  GFR between 60 and 89ml/min/1.73 m² / GFR between 15 and 29ml/min/1.73 m² / GFR < 15 ml/min/1.73 m²
Presence of other complications: dialysis | Day 0
  YES/NO
Presence of other complications: dialysis | Month 12
  YES/NO
Presence of other complications: dialysis | Month 24
  YES/NO
Presence of other complications: peripheral neuropathy | Day 0
  YES/NO and the nature thereof: monofilament (normal, pathological, not done)
Presence of other complications: peripheral neuropathy | Month 12
  YES/NO and the nature thereof: monofilament (normal, pathological, not done)
Presence of other complications: peripheral neuropathy | Month 24
  YES/NO and the nature thereof: monofilament (normal, pathological, not done)
Presence of other complications: vegetative neuropathy | Day 0
  YES/NO and the nature thereof: (bladder, digestive, erectile dysfunction, orthostatic arterial hypotension)
Presence of other complications: vegetative neuropathy | Month 12
  YES/NO and the nature thereof: (bladder, digestive, erectile dysfunction, orthostatic arterial hypotension)
Presence of other complications: vegetative neuropathy | Month 24
  YES/NO and the nature thereof: (bladder, digestive, erectile dysfunction, orthostatic arterial hypotension)
Presence of other complications: coronaropathy | Day 0
  YES/NO
Presence of other complications: coronaropathy | Month 12
  YES/NO
Presence of other complications: coronaropathy | Month 24
  YES/NO
Presence of other complications: heart failure | Day 0
  YES/NO
Presence of other complications: heart failure | Month 12
  YES/NO
Presence of other complications: heart failure | Month 24
  YES/NO
Presence of other complications: arteriopathy of the lower limbs | Day 0
  YES/NO and the nature thereof (revascularised or not/left or right side)
Presence of other complications: arteriopathy of the lower limbs | Month 12
  YES/NO and the nature thereof (revascularised or not/left or right side)
Presence of other complications: arteriopathy of the lower limbs | Month 24
  YES/NO and the nature thereof (revascularised or not/left or right side)
Presence of other complications: involvement of the supra-aortic trunk | Day 0
  YES/NO
Presence of other complications: involvement of the supra-aortic trunk | Month 12
  YES/NO
Presence of other complications: involvement of the supra-aortic trunk | Month 24
  YES/NO
Presence of other complications: stroke | Day 0
  YES/NO
Presence of other complications: stroke | Month 12
  YES/NO
Presence of other complications: stroke | Month 24
  YES/NO
Presence of other complications: sequellar hemiplegia | Day 0
  YES/NO
Presence of other complications: sequellar hemiplegia | Month 12
  YES/NO
Presence of other complications: sequellar hemiplegia | Month 24
  YES/NO
Treatments: oral antidiabetics | Day 0
  The nature of all oral antidiabetics will be recorded.
Treatments: oral antidiabetics | Month 12
  The nature of all oral antidiabetics will be recorded.
Treatments: oral antidiabetics | Month 24
  The nature of all oral antidiabetics will be recorded.
Treatments: injectable antidiabetics | Day 0
  The nature of all injectable antidiabetics will be recorded.
Treatments: injectable antidiabetics | Month 12
  The nature of all injectable antidiabetics will be recorded.
Treatments: injectable antidiabetics | Month 24
  The nature of all injectable antidiabetics will be recorded.
Other treatments | Day 0
  The nature of all other treatments will be recorded.
Other treatments | Month 12
  The nature of all other treatments will be recorded.
Other treatments | Month 24
  The nature of all other treatments will be recorded.
History of trophic disorders | Day 0
  YES/NO and, if so, left/right, both feet.
History of trophic disorders | Month 12
  YES/NO and, if so, left/right, both feet.
History of trophic disorders | Month 24
  YES/NO and, if so, left/right, both feet.
Regular pedicure treatments | Day 0
  The number and frequency of pedicure sessions per year will be recorded (if any).
Regular pedicure treatments | Month 12
  The number and frequency of pedicure sessions per year will be recorded (if any).
Regular pedicure treatments | Month 24
  YES/NO and, if so, number and frequency of pedicure sessions per year will be recorded (if any).
Weight | Day 0
  Kilos
Weight | Month 12
  Kilos
Weight | Month 24
  Kilos
Height | Day 0
  Centimeters
Height | Month 12
  Centimeters
Height | Month 24
  Centimeters
Charcot foot | Day 0
  Left/right/both
Charcot foot | Month 12
  Left/right/both
Charcot foot | Month 24
  Left/right/both
Estimated age of lesions (deformities) caused by neurogenic osteoarthropathy | Day 0
  In years
Estimated age of lesions (deformities) caused by neurogenic osteoarthropathy | Month 12
  In years
Estimated age of lesions (deformities) caused by neurogenic osteoarthropathy | Month 24
  In years
Neurogenic osteoarthropathy Sanders classification | Day 0
  Sanders 1: interphalangeal and metatarsophalangeal joints Sanders 2: tarsometatarsal joints Sanders 3 : naviculocuneiform, talonavicular or calcaneocuboid joints Sanders 4 : ankle joint, subtalar joint Sanders 5: calcaneum
Neurogenic osteoarthropathy Sanders classification | Month 12
  Sanders 1: interphalangeal and metatarsophalangeal joints Sanders 2: tarsometatarsal joints Sanders 3 : naviculocuneiform, talonavicular or calcaneocuboid joints Sanders 4 : ankle joint, subtalar joint Sanders 5: calcaneum
Neurogenic osteoarthropathy Sanders classification | Month 24
  Sanders 1: interphalangeal and metatarsophalangeal joints Sanders 2: tarsometatarsal joints Sanders 3 : naviculocuneiform, talonavicular or calcaneocuboid joints Sanders 4 : ankle joint, subtalar joint Sanders 5: calcaneum
Current mode of shoeing/unfastening at home | Day 0
  Barefoot and/or socks; serial sock; serial medical sock; normal shoe; normal medical shoe; foot orthosis; orthopedic low shaft shoe; orthopedic high shaft shoe; standard off-loading shoe; custom off-loading shoe ; standard removable boot; custom removable boot; non-removable boot; other...
Current mode of shoeing/unfastening outdoors | Day 0
  Barefoot and/or socks; serial sock; serial medical sock; normal shoe; normal medical shoe; foot orthosis; orthopedic low shaft shoe; orthopedic high shaft shoe; standard off-loading shoe; custom off-loading shoe ; standard removable boot; custom removable boot; non-removable boot; other...
Current mode of shoeing/unfastening at home | Month 12
  Barefoot and/or socks; serial sock; serial medical sock; normal shoe; normal medical shoe; foot orthosis; orthopedic low shaft shoe; orthopedic high shaft shoe; standard off-loading shoe; custom off-loading shoe ; standard removable boot; custom removable boot; non-removable boot; other...
Current mode of shoeing/unfastening outdoors | Month 12
  Barefoot and/or socks; serial sock; serial medical sock; normal shoe; normal medical shoe; foot orthosis; orthopedic low shaft shoe; orthopedic high shaft shoe; standard off-loading shoe; custom off-loading shoe ; standard removable boot; custom removable boot; non-removable boot; other...
Current mode of shoeing/unfastening at home | Month 24
  Barefoot and/or socks; serial sock; serial medical sock; normal shoe; normal medical shoe; foot orthosis; orthopedic low shaft shoe; orthopedic high shaft shoe; standard off-loading shoe; custom off-loading shoe ; standard removable boot; custom removable boot; non-removable boot; other...
Current mode of shoeing/unfastening outdoors | Month 24
  Barefoot and/or socks; serial sock; serial medical sock; normal shoe; normal medical shoe; foot orthosis; orthopedic low shaft shoe; orthopedic high shaft shoe; standard off-loading shoe; custom off-loading shoe ; standard removable boot; custom removable boot; non-removable boot; other...
Adherence to shoeing method | Day 0
  At home/outdoors
Adherence to shoeing method | Month 12
  At home/outdoors
Adherence to shoeing method | Month 24
  At home/outdoors
Presence of another trophic foot disorder during the previous year | Day 0
  YES/NO and date of onset of the ulcer (month and year)
Presence of another trophic foot disorder during the previous year | Month 12
  YES/NO and date of onset of the ulcer (month and year)
Presence of another trophic foot disorder during the previous year | Month 24
  YES/NO and date of onset of the ulcer (month and year)
Presence of a clinical infection | Day 0
  YES/NO and, if so, the Infectious Diseases Society of America classification
Presence of a clinical infection | Month 12
  YES/NO and, if so, the Infectious Diseases Society of America classification
Presence of a clinical infection | Month 24
  YES/NO and, if so, the Infectious Diseases Society of America classification
Foot or leg surgery in the previous year | Day 0
  YES/NO and, if so, left/right
Foot or leg surgery in the previous year | Month 12
  YES/NO and, if so, left/right
Foot or leg surgery in the previous year | Month 24
  YES/NO and, if so, left/right
Partial foot amputation | Day 0
  YES/NO and, if so, left/right
Partial foot amputation | Month 12
  YES/NO and, if so, left/right
Partial foot amputation | Month 24
  YES/NO and, if so, left/right
Trans-tibial amputation | Day 0
  YES/NO and, if so, left/right
Trans-tibial amputation | Month 12
  YES/NO and, if so, left/right
Trans-tibial amputation | Month 24
  YES/NO and, if so, left/right
Trans-femoral amputation | Day 0
  YES/NO and, if so, left/right
Trans-femoral amputation | Month 12
  YES/NO and, if so, left/right
Trans-femoral amputation | Month 24
  YES/NO and, if so, left/right
Other type of surgery | Day 0
  All other types of surgery : septic surgery / correction of morphostatic disorders of the forefoot / internal and/or external fixators / bone graft / correction of club foot will be recorded.
Other type of surgery | Month 12
  All other types of surgery : septic surgery / correction of morphostatic disorders of the forefoot / internal and/or external fixators / bone graft / correction of club foot will be recorded.
Other type of surgery | Month 24
  All other types of surgery : septic surgery / correction of morphostatic disorders of the forefoot / internal and/or external fixators / bone graft / correction of club foot will be recorded.
Hospitalization in the previous year | Day 0
  YES/NO and, if so, the reason why
Hospitalization in the previous year | Month 12
  YES/NO and, if so, the reason why
Hospitalization in the previous year | Month 24
  YES/NO and, if so, the reason why
Onset and management of a foot wound (medical or surgical) | Day 0
  YES/NO and dates
Onset and management of a foot wound (medical or surgical) | Month 12
  YES/NO and dates
Onset and management of a foot wound (medical or surgical) | Month 24
  YES/NO and dates
Management of a Charcot foot | Day 0
  YES/NO
Management of a Charcot foot | Month 12
  YES/NO
Management of a Charcot foot | Month 24
  YES/NO
Onset of a controlateral Charcot foot | Day 0
  YES/NO
Onset of a controlateral Charcot foot | Month 12
  YES/NO
Onset of a controlateral Charcot foot | Month 24
  YES/NO
Diabetic imbalance | Day 0
  YES/NO
Diabetic imbalance | Month 12
  YES/NO
Diabetic imbalance | Month 24
  YES/NO
Other comorbidity or other reason for surgery | Day 0
  YES/NO
Other comorbidity or other reason for surgery | Month 12
  YES/NO
Other comorbidity or other reason for surgery | Month 24
  YES/NO
Monitoring of glycemic control by HbA1c | Day 0
  HbA1c will be measured as a percentage
Monitoring of glycemic control by HbA1c | Month 12
  HbA1c will be measured as a percentage
Monitoring of glycemic control by HbA1c | Month 24
  HbA1c will be measured as a percentage
Monitoring of glomerular Filtration Rate | Day 0
  ml/mn
Monitoring of glomerular Filtration Rate | Month 12
  ml/mn
Monitoring of glomerular Filtration Rate | Month 24
  ml/mn
X-ray of Charcot foot under loading (profile view) | Day 0
  Measurement of the Djian Annonier angle and the Meary-Tomeno line
X-ray of Charcot foot under loading (profile view) | Month 12
  Measurement of the Djian Annonier angle and the Meary-Tomeno line
X-ray of Charcot foot under loading (profile view) | Month 24
  Measurement of the Djian Annonier angle and the Meary-Tomeno line
Front view X-ray of the ankle(s) under loading | Day 0
  With Meary cerclage (metal cerclage of the hindfoot)
Front view X-ray of the ankle(s) under loading | Month 12
  With Meary cerclage (metal cerclage of the hindfoot)
Front view X-ray of the ankle(s) under loading | Month 24
  With Meary cerclage (metal cerclage of the hindfoot)

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Centre Hospitalier de Boulogne-sur-Mer, Boulogne-sur-Mer, Pas-de-Calais
  - Groupement Hospitalier Est, Hôpital Cardiologique Service de Diabétologie 28 Av du Doyen Lépine, Bron
  - CH Sud Francilien Service de Diabétologie 40 Avenue Serge Dassault, Corbeil-Essonnes
  - CHU de Grenoble Service d'Endocrinologie Allée des Sablons Les écrins, Grenoble
  - Hôpital Hôtel dieu Service d'Endocrinologie 26 rue d'Harfleur, Le Creusot
  - CHU Bicêtre Service d'Endocrinologie et Maladies de la reproduction 78 rue du Général Leclerc, Le Kremlin-Bicêtre
  - CH de Lens Unité de Diabétologie-Endocrinologie- Nutrition-Obésité Centre Hospitalier Dr SCHAFFNER 99 rte de La Bassée,, Lens
  - CHRU de Lille Service d'Endocrinologie Diabétologie et Métabolisme, Hôpital Claude Huriez, Rue Polonovski, Lille
  - CHU de la CONCEPTION Service de Nutrition, Diabétologie, Obésité médicale, chirurgicale 47 Bd Baille, Marseille
  - CHU de Montpellier Service des Maladies métaboliques 371 av. Doyen Giraud, Montpellier
  - GH Pitié Salpétrière Unité de podologie Service de Diabétologie 47-83 Bd de l'Hôpital, Paris
  - GH Paris Saint Joseph Service de Diabétologie et Endocrinologie 185 rue Raymond Losserand, Paris
  - Hôpital Cochin Service de diabétologie 123 Bd de Port Royal, Paris
  - CHU de Lyon Sud Service d'Endocrinologie-Diabète-Nutrition CH Lyon Sud Pavillon médical, Bat 1B 165 chemin du Grand Revoyet, Pierre-Bénite
  - CHU Reims Service d'Endocrinologie, diabète-nutrition Rue du Général Koenig, Reims
  - Hôpitaux Universitaires de Strasbourg Service d'Endocrinologie et Diabétologie 1, place de l'hôpital,, Strasbourg
  - Hôpital DRON Service de diabétologie 135 rue du Président Coty, Tourcoing